CLINICAL TRIAL: NCT00658268
Title: Bisphosphonates and Impaction Grafting in Hip Revision Evaluated With Radiostereophotogrametri. A Randomized, Double-blind Study in Patients Operated for Aseptic Loosening and Osteolysis.
Brief Title: Bisphosphonates and Impaction Grafting in Hip Revision
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKOISR10001; EudraCT2006-006439-39
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Aseptic Loosening of the Hip Prosthesis
Keywords: Surgical procedures operative; Prosthesis implantation; Arthroplasty replacement
MeSH Terms: interventions — Clodronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Clodronate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clodronate — 60 mg/ml, 10 ml, single dose mixed in bone graft at operation
  Arms: 1
Drug: Placebo — 10 ml, single dose mixed in bone graft at operation
  Arms: 2

SUMMARY:
The primary focus of this study is to investigate whether increased bone density of the graft in revision arthroplasty of the hip can cause a decreased micromotion of the implant relative to the femur.

DETAILED DESCRIPTION:
Morsellized compacted bone allograft can be used for revision arthroplasty of the hip. Treating the graft locally with an antiresorptive substance such as a bisphosphonate has decreased the graft resorption in animal studies and led to a remained bone density in a human series of 16 patients. In the present study we investigate if this increased bone density of the graft also causes a decreased micromotion of the implant relative the femur. 36 patients are planned to participate in a 1:1 randomized and prospective study comparing the bisphosphonate Clodronate to saline. Primary outcome will be micromotion over the first year but also secondary parameters such as late micromotion (between 12 and 24 months), re-loosening subjective outcome and safety.

We hypothesize that rinsing the graft in a bisphosphonate solution prevents its resorption and therefore may reduce the risk of mechanical failure. Patients are followed with radiograms, RSA (radiostereography) preop, postop, at 6 weeks, at 12 and 24 months and subjective months and subjective parameters including Womac and SF 12. The treatment is simple, cheap and appears virtually risk-free.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aseptic loosening and osteolysis scheduled for hip revision using allograft and impaction technique
* Obtained informed consent
* Pregnancy excluded in women of childbearing age

Exclusion Criteria:

* Patients with known renal disease or S-creatinine >175 mcmol/L
* Patients with S-calcium 2.75 mmol/L
* Patients with diagnosed Rheumatoid arthritis
* Patients with active primary hyperparathyroidism

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Decrease of prosthetic micromotion from 2.7 mm to 1.7 mm as measured by RSA (0-24 months) | 12 months

SECONDARY OUTCOMES:
Decrease of prosthetic micromotion from 2.7 mm to 1.7 mm as measured by RSA (late micromotion) | 12-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Tagil, MD, PhD, Principal Investigator — Department of Orthopaedics, Lund University Hospital,Lund, Sweden
Locations (1):
- Lund University Hospital, Lund, Sweden